CLINICAL TRIAL: NCT00314444
Title: Treatment for Psychogenic Movement Disorders
Brief Title: Treatment for Psychogenic Disorders
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 060139; 06-N-0139
Record Dates: First submitted 2006-04-12; First posted 2006-04-13 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2009-04-14

CONDITIONS: Movement Disorders
Keywords: Psychogenic; Psychogenic Movement Disorders
MeSH Terms: conditions — Movement Disorders

SUMMARY:
This study will examine whether biofeedback treatment is effective in lessening or stopping movement symptoms in people with psychogenic movement disorder. People with this condition have increased or decreased movements that are not under their control and are not associated with any know problem with the nervous system. Biofeedback is a type of therapy that uses electronic instruments to monitor breathing and heart rate. This treatment has been effective in patients with anxiety and panic attacks.

People 18 years of age and older diagnosed with psychogenic movement disorder may be eligible for this study. Candidates are screened with a neurological history, physical examination and psychiatric evaluation.

Participants come to the NIH Clinical Center for nine 1-hour test sessions over an 8-week period for the following procedures:

Week 1 (two visits):

* Patients' movements are videotaped while they sit, stand and walk.
* Patients train on RESPeRATE device, a computerized musical biofeedback device to help slow theirs breathing rate. The device has three components: a computerized module, earphones, and a chest strap holding a breath sensor. The patients put the elastic strap around their chest, put on the earphones, and sit in a chair. The device monitors and analyzes their breathing to create a melody composed of two distinct tones - one for inhalation and one for exhalation. Patients are instructed to match their breathing to the tones, which gradually slow until they are breathing at a slower, therapeutic rate.
* Patients' breathing is monitored and analyzed for information on breathing pattern and rate.
* Patients complete questionnaires on level of relaxation before and after RESPeRATE training.
* Patients take the RESPeRATE device home to use for two 10-minute practice sessions per day. They complete relaxation questionnaires before and after each session.

Weeks 2-7:

* Patients' progress is monitored and reviewed from the previous week
* Patients' breathing is monitored and analyzed for information on breathing pattern and rate.
* Patients complete questionnaires on level of relaxation before and after RESPeRATE training.
* Patients are observed for 10 minutes while using the RESPeRATE device.

Week 8:

* Patients' progress is monitored and reviewed from the previous week
* Patients' breathing is monitored and analyzed for information on breathing pattern and rate.
* Patients complete questionnaires on level o...

DETAILED DESCRIPTION:
Objective:

To apply respiratory biofeedback to patients with Psychogenic Movement Disorders (PMD) with a goal of decreasing involuntary movements.

Study Population:

Patients diagnosed with "clinically definite" PMD based on the Fahn-Williams scale

Design: Open-label pilot study

Outcome measures:

* To evaluate a possible decrease or resolution in involuntary movements caused by PMD as measured by the Psychogenic Movement Disorder Scale. Videotaping will be performed pre- and post-treatment and the videos will be evaluated by movement disorder specialists who are blinded to the pre-treatment or post-treatment condition.
* To evaluate if respiratory biofeedback is an effective treatment for patients with PMD.
* To retrospectively evaluate the components of anxiety and depression with responders versus non-responders.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Clinically definite functional (psychogenic) movement disorder as defined by Fahn and Williams criteria diagnosed by a movement disorder neurologist.
* Patients who are at least 18 years old
* Able and willing to cooperate with the study requirements

EXCLUSION CRITERIA:

* Any underlying major medical or neurological conditions
* Patients whose movements are related to a known neurological disorder
* History of traumatic brain injury or history of strokes
* Current suicidal ideation
* Patients with a psychotic disorder
* Patients with active substance abuse within the last 6 months
* Patients with moderate to severe depression, Beck Depression Inventory (BDI) greater than 18)
* Patients with any ongoing litigation related to their diagnosis of PMD.
* Patients with a definite overt stressor identified that is thought to be primarily responsible for the PMD symptoms

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15
Dates: Start 2006-04-07; Study Completion 2009-04-14

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Thomas M, Jankovic J. Psychogenic movement disorders: diagnosis and management. CNS Drugs. 2004;18(7):437-52. doi: 10.2165/00023210-200418070-00003. PMID 15139799
- [Background] Factor SA, Podskalny GD, Molho ES. Psychogenic movement disorders: frequency, clinical profile, and characteristics. J Neurol Neurosurg Psychiatry. 1995 Oct;59(4):406-12. doi: 10.1136/jnnp.59.4.406. PMID 7561921
- [Background] Anderson KE. Psychogenic Movement Disorders. Curr Treat Options Neurol. 2003 Mar;5(2):169-176. doi: 10.1007/s11940-003-0007-y. PMID 12628065